CLINICAL TRIAL: NCT06760897
Title: The Clinical Efficacy Study of Selective Gastrogenic Microbiota Transplantation in the Treatment of Functional Dyspepsia
Brief Title: Effect of Gastrogenic Microbiota in FD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFEC-2024-670
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Dyspepsia; Dysbiosis
MeSH Terms: conditions — Dyspepsia; Dysbiosis

STUDY DESIGN:
Intervention Model Description: randomized placebo-controlled study in 2 parallel FD cohorts
Who Masked: Participant, Care Provider, Investigator
Masking Description: participants, care providers, and investigators are blinded during the randomized placebo-controlled phase (8 weeks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cohort 1FD (Experimental): Receiving 8 weeks of Gastrogenic Microbiota
  Interventions: Dietary Supplement: Gastrogenic Microbiota
- cohort 2FD (Placebo Comparator): Receiving 8 weeks of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Gastrogenic Microbiota — Take 1 sachet of gastric-origin probiotic powder (containing 5 x 1011 CFU per sachet) twice daily for 8 weeks.
  Arms: cohort 1FD
Other: Placebo — similar powder administered twice daily
  Arms: cohort 2FD

SUMMARY:
Single-center prospective interventional study aimed at demonstrating the effect of gastric-origin probiotics on dyspeptic symptoms, tryptophan metabolism, and microbiome parameters in FD patients without Helicobacter pylori infection, compared to a placebo group

DETAILED DESCRIPTION:
Prospective randomized placebo-controlled study in 2 parallel FD cohorts (8 weeks) :

cohort 1FD : Receiving 8 weeks of Gastrogenic Microbiota cohort 2FD : Receiving 8 weeks of placebo Clinical outcomes and Tryptophan metabolism, Microbiome parameters will be assessed at the beginning and end of each treatment period (week 0, 8).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 and ≤70 years, with symptoms such as upper abdominal pain or burning sensation, postprandial bloating, early satiety, etc., and who meet the diagnostic criteria for functional dyspepsia (FD) according to the Rome IV criteria.
* Negative result on the C13 urea breath test, and no organic changes observed on gastroscopy.

Exclusion Criteria:

* Use of acid-suppressing drugs, prokinetic agents, antibiotic or anxiolytics within 4 weeks prior to enrollment.
* History of abdominal surgery, abdominal or inflammatory bowel disease, diabetes, active psychiatric disorders, or severe diseases of vital organs such as the heart, lungs, liver, or kidneys.
* Pregnant or breastfeeding participants, or those currently involved in other clinical research studies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
The rate of relief of functional dyspepsia symptoms in Lactobacillus vs. placebo | 8 weeks
  The rate of relief of functional dyspepsia symptoms in Lactobacillus vs. placebo [Time Frame: 8 weeks] (using the the Patient Assessment of Upper Gastrointestinal Symptom Severity Index PAGI-SYM).The PAGI-SYM scale is specifically developed for the assessment of functional upper gastrointestinal diseases and is used to evaluate the severity of symptoms associated with these diseases. The scale comprises 21 symptoms of functional upper gastrointestinal diseases, with each symptom rated on a scale from none to very severe, scored as 0, 1, 2, 3, 4, or 5, respectively. The total score is calculated and used to assess the severity of functional upper gastrointestinal diseases.

SECONDARY OUTCOMES:
Changes in the Clinical Rating Scale for The Gastrointestinal Symptoms Rating Scale (GSRS) scores in the Lactobacillus vs. the placebo. | 8 weeks
  The Gastrointestinal Symptom Rating Scale (GSRS) is specifically designed for the assessment of gastrointestinal symptoms, particularly in patients with gastroesophageal reflux disease. This scale consists of a series of questions aimed at evaluating the severity of various gastrointestinal symptoms experienced by the patient over the past week. The GSRS includes items such as pain or discomfort in the upper abdomen, heartburn, and acid reflux, each rated on a scale from 'no discomfort at all' to 'very severe discomfort'. The ratings are scored on a seven-point Likert scale, ranging from 0 to 6, with higher scores indicating more severe symptoms. The total score is calculated by summing the scores of all items, providing a comprehensive assessment of the patient's gastrointestinal symptom severity.
Changes in the Quality of Life scores (PAGI-QOL) in the Lactobacillus vs. the placebo. | 8 weeks
  The Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) is specifically designed to assess the quality of life in patients with upper gastrointestinal disorders, including dyspepsia, gastroesophageal reflux disease (GERD), and gastroparesis. This questionnaire consists of 30 items covering five domains: Daily Activities, Clothing, Diet and Food Habits, Relationship, and Psychological Well-Being and Distress. Each item is scored to reflect the impact of the disorder on the patient's quality of life, with higher scores indicating a greater impact. The PAGI-QOL has demonstrated excellent internal consistency, with a Cronbach's alpha ranging from 0.83 to 0.96, ensuring its reliability and validity in assessing the quality of life in these patients.
Changes in the Self-Rating Anxiety Scale (SAS) scores in the Lactobacillus vs. the placebo. | 8 weeks
  The Self-Rating Anxiety Scale (SAS) is a widely-used psychological assessment tool, developed by Dr. William W. K. Zung, specifically designed to quantify the level of anxiety in individuals. The SAS is structured to assess various dimensions of anxiety, including cognitive, affective, somatic, and autonomic symptoms, providing a comprehensive overview of an individual's anxiety level. This scale consists of 20 items, each scored on a four-point scale ranging from 1 (none or some of the time) to 4 (most or all of the time), with a total score ranging from 20 to 80, with higher scores indicating more severe anxiety symptoms. The items are phrased to reflect common experiences of people with anxiety, making it a practical tool for both clinical and research settings. It is primarily used to evaluate the presence and intensity of anxiety symptoms, serving as a valuable instrument in the assessment and monitoring of anxiety disorders.
Changes in the Self-Rating Depression Scale (SDS) scores in the Lactobacillus vs. the placebo. | 8 weeks
  The Self-Rating Depression Scale (SDS) is a widely-used psychological assessment tool developed by Dr. William W. K. Zung, designed to measure the presence and severity of depressive symptoms in individuals. This scale consists of 20 items, each assigned a rating on a scale from 1 (none or some of the time) to 4 (most or all of the time), with a total score ranging from 20 to 80, with higher scores indicating more severe depressive symptoms. The SDS is designed to measure the affective, psychological, and somatic aspects of depression, enabling clinicians to better understand and diagnose the condition in their patients. The SDS is a valuable tool in clinical and research settings for assessing depression and its associated factors across diverse populations. Its simple structure and straightforward administration make it an accessible and effective method for measuring depressive symptoms.
Differences in the composition of gastric mucosal and fecal microbiota before and after treatment in the probiotic group | 8 weeks
  Differences in the composition of gastric mucosal and fecal microbiota before and after treatment in the probiotic group
Differences in serum and urine neurotransmitters before and after treatment in the probiotic group | 8 weeks
  Differences in serum and urine neurotransmitters before and after treatment in the probiotic group
Safety of Lactobacillus vs. placebo | 8 weeks
  number of adverse events with sporebiotics vs. placebo

CONTACTS AND LOCATIONS:
Locations (1):
- NanfangH, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No